CLINICAL TRIAL: NCT01122537
Title: Clinical Features, Microbiological Characteristics, and Differential Diagnosis of Postneurosurgical Meningitis
Brief Title: Characterization and Differential Diagnosis of Postneurosurgical Meningitis
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-Ho Choi, Doctor, Asan Medical Center
Other Study IDs: APNSM
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Neurosurgery
Keywords: Meningitis; infection; cerebrospinal fluid; procalcitonin; adenosine deaminase
MeSH Terms: conditions — Meningitis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Meningitis is a rare complication following neurosurgical procedures and is associated with high morbidity and mortality. The aim of this study is to describe the clinical characteristics and microbiological characteristics in patients who develope meningitis following neurosurgical operations, and investigate the useful tips for the differential diagnosis of postneurosurgical meningitis.

DETAILED DESCRIPTION:
Besides description of characteristics of patients with postneurosurgical patients, we also will investigate the usefulness of prolonged cerebrospinal fluid (CSF) culture, and profiles of blood and CSF inflammatory markers for the differential diagnosis of meningitis. CSF culture will be extended upto 2 weeks. Serum procalcitonin and C-reactive protein, CSF adenosine deaminase levels will be monitored and analyzed for the differential diagnosis of meningitis.

ELIGIBILITY:
Inclusion Criteria:

* Cerebrospinal fluid corrected WBC >6/mm^3 and/or fever (> 38℃) and/or neck stiffness

Exclusion Criteria:

* Patients already treated more than 48 hours for meningitis before cerebrospinal fluid examination

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient who develop meningitis after neurosurgical operation
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Development of meningitis | within 4 weeks after neurosurgical operation

SECONDARY OUTCOMES:
All-cause mortality | within 4 weeks after the diagnosis of meningitis

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ho Choi, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea